CLINICAL TRIAL: NCT06580509
Title: TranExamic Atomized for Pediatric Post-Operative Tonsillectomy Hemorrhage (TEAPOT): A Pilot and Feasibility Study
Brief Title: TranExamic Atomized for Pediatric Post-Operative Tonsillectomy Hemorrhage: Pilot Study
Acronym: TEAPOT
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000638
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhage, Surgical; Tonsillar Bleeding
Keywords: Tranexamic Acid; Nebulizer; Post tonsillectomy hemorrhabe
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Two arm randomized, double-blind, controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: To maintain blinding, all personnel except the investigational pharmacist and/or statistician will be unaware of the administered drug.
  The randomization schedule will be pre-determined by a central randomization process and prepared as "use next boxes" to streamline the process at enrollment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nebulized Tranexamic Acid (Experimental): Subjects will be adminstered nebulized TXA post-tonsillectomy if they return to the emergency room with hemorrhage after surgery
  Interventions: Drug: Tranexamic Acid Injectable Product
- Nebulized Saline (Placebo Comparator): Subjects will be adminstered nebulized saline post-tonsillectomy if they return to the emergency room with hemorrhage after surgery
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Tranexamic Acid Injectable Product — Participants will receive three doses of TXA 500 mg (5 mL of TXA 100mg/ml) nebulized using a PARI LC D Disposable Nebulizer or equivalent over 10-15 minutes using 8 or greater liter/minute of gas flow.
  Other Names: TXA 100mg/ml
  Arms: Nebulized Tranexamic Acid
Other: Normal Saline — Participants will receive three 5 ml doses of placebo (normal saline) nebulized using a PARI LC D Disposable Nebulizer or equivalent over 10-15 minutes using 8 or greater liter/minute of gas flow.
  Other Names: 0.9% saline solution
  Arms: Nebulized Saline

SUMMARY:
After a child has their tonsils removed, sometimes they might bleed which can be a problem. There is a special mist medicine called nebulized tranexamic acid (TXA) that might help stop the bleeding without having to touch the sore spot. If this mist works well, it could help kids get better by making sure they don't have to go back for more surgery or need blood from someone else. Not having another surgery is good because it means kids won't have to sleep under medicine again, which can sometimes be risky for their brains and breathing, and they won't feel as scared or hurt.

DETAILED DESCRIPTION:
The study intervention involves administering nebulized tranexamic acid (TXA) to pediatric patients with traumatic hemorrhage (PTH). The intervention consists of three consecutive doses of nebulized TXA.

The dosage of nebulized TXA is adjusted based on the child's weight. For children weighing more than 25 kg, each dose is 500 mg. For children weighing less than 25 kg, each dose is 250 mg.

Frequency: The three doses of nebulized TXA are administered consecutively over the course of approximately an hour. Administration Method: Nebulized TXA is delivered through a nebulizer device. A nebulizer converts the liquid medication into a fine mist or aerosol, which is then inhaled by the patient. This method allows the medication to be delivered directly to the respiratory tract, where it can exert its effect on the bleeding site. Delivery Setting: The intervention may take place in a clinical setting, such as a hospital or outpatient clinic, where nebulizer devices and medical supervision are readily available. Each patient receives three nebulized independent doses of TXA in succession. The delivery of the intervention is carried out by healthcare professionals trained in administering nebulized medications.

ELIGIBILITY:
Inclusion Criteria:

1. Received a tonsillectomy
2. Presents to the ED with secondary* post-tonsillectomy hemorrhage
3. Children between age of 2 to 17 years of age (i.e., before their 18th birthday) *Secondary post-tonsillectomy hemorrhage is defined as greater than 24 hours from their primary tonsillectomy operation (arrival in recovery/PACU).

Exclusion Criteria:

1. Known and documented bleeding or clotting disorder.
2. Known pregnancy.
3. Patients with known hypersensitivity or allergic response to tranexamic acid.
4. Parents or guardians who cannot communicate in English or Spanish.
5. Intubation prior to enrollment.
6. Previously enrolled patients.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled per month | Baseline to 18 months (or duration of study)
  Assess target enrollment of patients per site per month.
Number of nebulizations per patient | Baseline to 18 months (or duration of study)
  Evaluate the ability to nebulize at least two doses of TXA to children with PTH
Indirect local concentration of nebulized TXA | Immediately post nebulizer treatment (within 60 minutes) and then within 8 hours.
  Limited data on nebulized TXA systematic absorption. Topical PK studies of TXA document a significant reduction in systematic levels but the same hemostasis effect. Collection of two blood samples from each participant. This will verify a pulmonary physiological-based PK model (PBPK) (i.e., nasal cavity, pharynx, and lung) that indirectly predicts the oropharyngeal and systematic concentration of nebulized TXA.
Systemic Concentration of nebulized TXA | Immediately post nebulizer treatment (within 60 minutes) and up to eights hours.
  Pharmacokinetics samples will be collected after completion of the last nebulized treatment received within sixty minutes. A second time point should then be collected after sixty minutes up to eight hours from last nebulization, separated from the previous time point by at least sixty to ninety minutes. The serum TXA levels will be used to verify a TXA Physiological-based Pharmacokinetic model and determine the population variability. This PBPK model is built by our research pharmacist based on extensive research already completed on TXA distribution and metabolism. Once the model is built, the investigators only need a one to two samples to determine if the model accurately reflects collect samples. The investigators will develop a base model to determine a best-fit compartmental model, distribution, and elimination kinetics. The investigators will also use stochastic models to evaluate between-subject variability in PK parameters.

SECONDARY OUTCOMES:
Number of return visits to the OR | Baseline to 18 months (or duration of study)
  The need for return to the Operating Room (OR) for surgical management of PTH) will be followed for up to seven days after randomization
Estimated blood loss | Baseline to 7 days
  Determine the estimated blood loss per participant
Number of recurrences of PTH | Baseline to 18 months (or duration of study)
  Number of participants in which there was a recurrence of post-tonsillectomy hemorrhage after the study drug was administered
Number of blood transfusions required | Baseline to 18 months (or duration of study)
  Blood product transfusion volume will be measured at discharge or 24 hours (whichever comes first). This will include the volume of packed red blood cells, platelets, plasma, cryoprecipitate, or whole blood. Any mention of blood loss in electronic health records from emergency, anesthesiology, or surgeons' notes will be recorded.

OTHER OUTCOMES:
Wong-Baker FACES Pain Rating Scale | Day 1, 7 and 30
  The participant rates their pain from 0=No hurt to 10=Hurts worst
State-Trait Anxiety Inventory (STAI) for Adults | Day 1 and day 7 plus or minus one day.
  A widely used self-reported anxiety assessment instrument with versions for children over eight years of age, adolescents, and adults is the State-Trait Anxiety Inventory (STAI). The assessment is composed of two separate scales used in assessing situational (STAI-State) and baseline (STAI-Trait) anxiety levels. For more information please see https://www.mindgarden.com/145-state-trait-anxiety-inventory-for-adults.
  Scale Range: Each part (State and Trait) of the STAI consists of 20 items, with scores ranging from 20 to 80. State Anxiety: Reflects how the respondent feels at a particular moment (e.g., calm, tense). Trait Anxiety: Measures how the respondent generally feels over time (e.g., relaxed, nervous).
  Score Interpretation: Higher Scores: Indicate higher levels of anxiety. A score above 40 is generally considered to suggest significant anxiety symptoms.
  Lower Scores: Indicate lower levels of anxiety.
State-Trait Anxiety Inventory for Children (STAIC) | Day 1 and Day 7 (plus or minus one day)
  Scale Range: Similar to the adult version, the STAIC has separate scales for state and trait anxiety, each with 20 items. Scores range from 20 to 60 for each scale.
  State Anxiety: Measures how children feel at the moment. Trait Anxiety: Assesses how children usually feel over time.
  Score Interpretation: Higher Scores: Reflect higher levels of anxiety. A score above 30 on either scale may indicate elevated anxiety. Lower Scores: Suggest lower levels of anxiety.
  Interpretation: High State Anxiety Scores: Indicate a current feeling of anxiety or stress, possibly due to a specific situation or event. High Trait Anxiety Scores: Suggest a predisposition to experiencing anxiety more frequently or intensely over time. Low Scores (Both State and Trait): Indicate calmness and a lower likelihood of anxiety, whether temporarily or as a general tendency.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Meyer, MD, MS, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Hospital, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results in Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results in information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested by other researchers 3 years after the completion of the primary endpoint by contacting Andrew D. Meyer, MD, MS or through the DCC public use dataset website.